CLINICAL TRIAL: NCT06985290
Title: Comparative Efficacy of Dexmedetomidine Versus Morphine in Alleviating Secondary Brain Injury, When Used for Sedation During Hypothermia Therapy in Neonates: A Pilot Randomized Trial
Brief Title: Dexmedetomidine Versus Morphine During Cooling Therapy in Neonates
Acronym: COOL-SED
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsita Goswami (Other)
Responsible Party: Sponsor-Investigator, Ipsita Goswami, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20027280
Record Dates: First submitted 2025-03-27; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hypoxic Ischemic Brain Injury; Neonatal Encephalopathy; Perinatal Anoxic-ischemic Brain Injury
Keywords: sedation; analgesia; dexmedetomidine; morphine
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): Dexmedetomidine infusion as sedation during therapeutic hypothermia and rewarming
  Interventions: Drug: Dexmedetomidine Infusion
- Morphine Group (Active Comparator): Morphine infusion as sedative during therapeutic hypothermia and rewarming
  Interventions: Drug: Morphine Infusion

INTERVENTIONS:
Drug: Dexmedetomidine Infusion — Dexmedetomidine infusion given for sedation during therapeutic hypothermia. Dexmedetomidine infusion at a starting dose of 0.2 μg/kg/h, with titration in 0.1 μg/kg/h increments with a maximum of 0.5 μg/kg/h based on objective assessment of sedation.
  Arms: Dexmedetomidine Group
Drug: Morphine Infusion — Morphine infusion given for sedation during therapeutic hypothermia. Morphine infusion at a starting dose of 4 μg/kg/h, with titration in 2 μg/kg/h increments with a maximum of 10 μg/kg/h based on objective assessment of sedation.
  Arms: Morphine Group

SUMMARY:
About ~3/ 1000 live-born newborns may suffer from brain injury due to a transient drop in oxygen supply to the brain during the birth process. The degree of brain injury that ensues in the first 72 hours after the injury is directly proportional to the severity of long-term childhood disabilities (e.g., cerebral palsy and developmental delays). Whole-body cooling during the first 3 days of life is proven effective in reducing the severity of brain injury. However, cooling therapy leads to pain, shivering, stress, and discomfort. The best way to alleviate the pain and agitation of cooled newborns is unknown. Standard practice is to provide morphine infusion to reduce pain. Recently, a new drug called "dexmedetomidine" has been tested in small studies and has been found to be safe during cooling in newborns. Dexmedetomidine has added beneficial effects such as anti-inflammation, faster recovery, and shorter hospital stays. This study is going to test the feasibility of conducting a future clinical trial to compare the effects of using Dexmedetomidine versus morphine in the management of cooling-related pain/agitation on the severity of brain injury in the first week of life. The study will also examine the effect of dexmedetomidine compared to morphine on short-term clinical outcomes, parental experiences and developmental outcomes at 1 year.

ELIGIBILITY:
Inclusion criteria:

1. Gestational age >= 35 weeks
2. Birth weight >= 2500g
3. Sign of perinatal hypoxic event (any of the following): (a) Arterial Cord blood gas or postnatal gas within 1 hour of life pH <= 7.00 OR Base Deficit >= 16 (b) Arterial Cord blood gas postnatal gas within 1 hour of life pH 7.00 -7.15 AND Acute sentinel intrapartum event
4. Sign of Neonatal Encephalopathy
5. Initiation of Therapeutic Hypothermia within 8 hours of life

Exclusion criteria:

1. Informed consent not obtained within 20 hours of life
2. Congenital Brain Malformations (antenatally known)
3. Major Chromosomal Anomaly (antenatally diagnosed)
4. Congenital neuromuscular disorder

Max Age: 20 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Day 1
  Proportion of eligible neonates enrolled. Calculation = (Number of neonates enrolled) X 100/(Total eligible neonates)
Follow Up Rate | From enrollment to 1 year of age
  Percentage of neonates completing the study. Calculation = (Neonates who completed the study) x 100/ (Total neonates consented)
Adverse Event Rate | From enrollment to 7 days of life
  Incidence of adverse events Measurement of Adverse Event Rate = (Number of neonates experiencing) x100/ (Total neonates exposed to the intervention)
Discontinuation Rate | From enrollment to 7 days of life
  Need for intervention discontinuation due to adverse effects. Measurement of Discontinuation Rate = (Number of neonates for whom the intervention discontinued) x 100/ (Total neonates consented)
Protocol Adherence Rate | through study completion, average 1 year
  Percentage of correct drug adjustment based on changes in COMFORTneo scale as per protocol. Calculation of Drug Administration Compliance = (Number of correctly administered medication per month) x 100/ (Total number of participant enrolled per month)

SECONDARY OUTCOMES:
Severity of Brain Injury on Magnetic Resonance Imaging (MRI) | From enrollment to 10 days of life
  The T1 and T2 weighted images, diffusion-weighted images, and magnetic resonance spectroscopy (MRS) are additionally evaluated to determine the level of brain damage. MRI scoring system reported by Weeke et al. will be used to classify brain injury based on 4 subscores, including grey matter (basal ganglia, thalamus, PLIC, brainstem, perirolandic cortex, and hippocampus), white matter/cortex (including optic radiation and corpus callosum), and cerebellum.
Seizure Burden during Therapeutic Hypothermia | From enrollment to 72 hours of life
  Total duration of seizures noted during the first 72 hours of life
Stress levels measured by Salivary cortisol assay at 24 and 48 hours | From enrollment to 48 hours of life
  Salivary cortisol levels will be used as an objective marker of neonatal stress measured in µg/dL.
Neonatal Sedation and Discomfort Levels | From enrollment to 4 days of life
  COMFORT neo scores during the period of therapeutic hypothermia. It consists of 7 behavioural items (alertness, calmness/agitation, respiratory response, crying, body movement, facial tension and muscle tone), of which six items should be scored (respiratory response or crying depends on the presence of invasive ventilation). The neonate will be observed for 2 minutes to score. Total scores range from 7 to 35. A score >14 is considered a sign of distress and undersedation. A score < 9 suggests oversedation.
Time to Reach Full Oral Feeds | up to 4 weeks of life
  Days of life when participant is receiving all oral feeds either breast or bottle
Cumulative dose of PRN opioid boluses given during therapeutic hypothermia | up to 4 days of life
  Total dose of morphine and fentanyl given during therapeutic hypothermia measured in mg/kg of morphine equivalent
Length of Hospital Stay | up to 4 weeks of life
  Day of life when discharged home
Days on invasive and non-invasive respiratory support | Up to 4 weeks of life
  Day of life when comes off all respiratory support to room air

OTHER OUTCOMES:
Parental Stress Index | Up to 4 weeks of life
  Parental Stress Index - Short Form (PSI-SF) will be administered to parents of study subjects at discharge from NICU to compare stress levels between neonates of the two groups. The short form is derived from the original Parental Stress Index (PSI). It consists of 36 items across three subscales namely (i) Parental Distress (PD): stress related to personal factors (e.g., depression, lack of support), (ii) Parent-Child Dysfunctional Interaction (P-CDI): stress about the child not meeting expectations and (iii) Difficult Child (DC): stress due to child's behavioral difficulties. Each item is rated 1 (Strongly Disagree) to 5 (Strongly Agree). Percentiles based on normative data are used to interpret scores.
  >85th percentile indicates clinically significant stress, 90th-99th percentile indicates highly elevated stress.
Parental Experiences | From discharge to 4 weeks post-discharge
  Parental experiences captured through semi-structured interviews will be audio-recorded and transcribed.
Developmental Outcomes at 12 months | Between 10-14 months of enrollment
  Ages and Stages Questionnaire-3rd edition (ASQ-3) to assess five areas of childhood development: Communication, Gross motor, Fine motor, Problem-solving, and Personal-social through parent/caregiver reports. Each item is answered as Yes (10 points), Sometimes (5 points) and Not Yet (0 points).
  Each domain has 6 questions, hence a maximum 60 points per domain. After summing scores for each domain, total score is interpretated as: (i) Above Cutoff (Development is on schedule), (ii) Close to Cutoff (within 1 SD) (Monitor, Child may need re-screening soon) and (iii) Below Cutoff (Referral to specialist for further evaluation recommended).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsita Goswami, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with qualified researchers following publication of the primary study results. Data sharing will comply with applicable privacy regulations (e.g., PIPEDA/PHIPA).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available beginning 12 months after publication of the primary results or within 18 months of primary study completion, whichever occurs first. Data will be available for at least 5 years thereafter.
Access Criteria: Researchers must submit a scientifically sound proposal. Access will be granted upon approval by the Data Access Committee and signing of a Data Use Agreement (DUA). Data must be used for secondary analyses, meta-analyses, or validation studies. Re-identification attempts are prohibited.

REFERENCES:
- [Background] Alvik A, Groholt B. Examination of the cut-off scores determined by the Ages and Stages Questionnaire in a population-based sample of 6 month-old Norwegian infants. BMC Pediatr. 2011 Dec 19;11:117. doi: 10.1186/1471-2431-11-117. PMID 22182217
- [Background] Weeke LC, Groenendaal F, Mudigonda K, Blennow M, Lequin MH, Meiners LC, van Haastert IC, Benders MJ, Hallberg B, de Vries LS. A Novel Magnetic Resonance Imaging Score Predicts Neurodevelopmental Outcome After Perinatal Asphyxia and Therapeutic Hypothermia. J Pediatr. 2018 Jan;192:33-40.e2. doi: 10.1016/j.jpeds.2017.09.043. PMID 29246356
- [Background] Craig A, Deerwester K, Fox L, Jacobs J, Evans S. Maternal holding during therapeutic hypothermia for infants with neonatal encephalopathy is feasible. Acta Paediatr. 2019 Sep;108(9):1597-1602. doi: 10.1111/apa.14743. Epub 2019 Mar 5. PMID 30721531
- [Background] Meesters NJ, Dilles T, van Rosmalen J, van den Bosch GE, Simons SHP, van Dijk M. COMFORTneo scale: a reliable and valid instrument to measure prolonged pain in neonates? J Perinatol. 2023 May;43(5):595-600. doi: 10.1038/s41372-023-01628-1. Epub 2023 Feb 6. PMID 36746985
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Background] Elliott M, Fairchild K, Zanelli S, McPherson C, Vesoulis Z. Dexmedetomidine During Therapeutic Hypothermia: A Multicenter Quality Initiative. Hosp Pediatr. 2024 Jan 1;14(1):30-36. doi: 10.1542/hpeds.2023-007403. PMID 38115800
- [Background] McAdams RM, Pak D, Lalovic B, Phillips B, Shen DD. Dexmedetomidine Pharmacokinetics in Neonates with Hypoxic-Ischemic Encephalopathy Receiving Hypothermia. Anesthesiol Res Pract. 2020 Feb 25;2020:2582965. doi: 10.1155/2020/2582965. eCollection 2020. PMID 32158472
- [Background] Joshi M, Muneer J, Mbuagbaw L, Goswami I. Analgesia and sedation strategies in neonates undergoing whole-body therapeutic hypothermia: A scoping review. PLoS One. 2023 Dec 7;18(12):e0291170. doi: 10.1371/journal.pone.0291170. eCollection 2023. PMID 38060481
- [Background] Backe P, Bruschettini M, Blomqvist YT, Sibrecht G, Olsson E. Interventions for the Management of Pain and Sedation in Newborns Undergoing Therapeutic Hypothermia for Hypoxic-Ischemic Encephalopathy: A Systematic Review. Paediatr Drugs. 2023 Jan;25(1):27-41. doi: 10.1007/s40272-022-00546-7. Epub 2022 Dec 8. PMID 36481984
- [Background] Walker SM. Long-term effects of neonatal pain. Semin Fetal Neonatal Med. 2019 Aug;24(4):101005. doi: 10.1016/j.siny.2019.04.005. Epub 2019 Apr 5. PMID 30987942
- [Background] Wu Y, Kapse K, Jacobs M, Niforatos-Andescavage N, Donofrio MT, Krishnan A, Vezina G, Wessel D, du Plessis A, Limperopoulos C. Association of Maternal Psychological Distress With In Utero Brain Development in Fetuses With Congenital Heart Disease. JAMA Pediatr. 2020 Mar 1;174(3):e195316. doi: 10.1001/jamapediatrics.2019.5316. Epub 2020 Mar 2. PMID 31930365
- [Background] Thoresen M, Satas S, Loberg EM, Whitelaw A, Acolet D, Lindgren C, Penrice J, Robertson N, Haug E, Steen PA. Twenty-four hours of mild hypothermia in unsedated newborn pigs starting after a severe global hypoxic-ischemic insult is not neuroprotective. Pediatr Res. 2001 Sep;50(3):405-11. doi: 10.1203/00006450-200109000-00017. PMID 11518829
- [Background] van Marken Lichtenbelt WD, Schrauwen P. Implications of nonshivering thermogenesis for energy balance regulation in humans. Am J Physiol Regul Integr Comp Physiol. 2011 Aug;301(2):R285-96. doi: 10.1152/ajpregu.00652.2010. Epub 2011 Apr 13. PMID 21490370
- [Background] Mohammad K, McIntosh S, Lee KS, Beltempo M, Afifi J, Tremblay S, Shah P, Wilson D, Bodani J, Khurshid F, Makary H, Ng E, Wintermark P; NeoBrainNetwork. Variations in care of neonates during therapeutic hypothermia: call for care practice bundle implementation. Pediatr Res. 2023 Jul;94(1):321-330. doi: 10.1038/s41390-022-02453-6. Epub 2023 Jan 9. PMID 36624286
- [Background] Goswami IR, Whyte H, Wintermark P, Mohammad K, Shivananda S, Louis D, Yoon EW, Shah PS; Canadian Neonatal Network Investigators. Characteristics and short-term outcomes of neonates with mild hypoxic-ischemic encephalopathy treated with hypothermia. J Perinatol. 2020 Feb;40(2):275-283. doi: 10.1038/s41372-019-0551-2. Epub 2019 Nov 13. PMID 31723237
- [Background] Jacobs SE, Berg M, Hunt R, Tarnow-Mordi WO, Inder TE, Davis PG. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003311. doi: 10.1002/14651858.CD003311.pub3. PMID 23440789
- [Background] Shankaran S. Therapeutic hypothermia for neonatal encephalopathy. Curr Treat Options Neurol. 2012 Dec;14(6):608-19. doi: 10.1007/s11940-012-0200-y. PMID 23007949
- [Background] Kromm GH, Patankar H, Nagalotimath S, Wong H, Austin T. Socioemotional and Psychological Outcomes of Hypoxic-Ischemic Encephalopathy: A Systematic Review. Pediatrics. 2024 Apr 1;153(4):e2023063399. doi: 10.1542/peds.2023-063399. PMID 38440801
- [Background] Pisani F, Orsini M, Braibanti S, Copioli C, Sisti L, Turco EC. Development of epilepsy in newborns with moderate hypoxic-ischemic encephalopathy and neonatal seizures. Brain Dev. 2009 Jan;31(1):64-8. doi: 10.1016/j.braindev.2008.04.001. Epub 2008 May 19. PMID 18490125